CLINICAL TRIAL: NCT05119361
Title: Impact on the Fluid Balance of a Perfusion Based Protocol to Adjust UFnet During Deresuscitation in Intensive Care Unit. A Before-after Study.
Brief Title: Early Dry Cohort : Impact on the Fluid Balance of a Perfusion Based Protocol to Adjust UFnet During Deresuscitation in Intensive Care Unit.
Acronym: Early Dry
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 454
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Acute Kidney Injury
Keywords: ultrafiltration; deresuscitation; fluid overload; fluid balance.
MeSH Terms: conditions — Acute Kidney Injury; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- before protocol implementation: A control group reflecting usual practice about net ultrafiltration and deresuscitation strategy in patients with continuous renal replacement therapy in our Department.
  All patients meeting eligibility criteria between 01/01/2020 and 31/12/2021 will be include.
  Interventions: Other: Early Dry protocol
- after protocol implementation: All patients treated by our deresuscitation protocol between 15/02/2020 and 15/08/2021 will be included.
  Interventions: Other: Early Dry protocol

INTERVENTIONS:
Other: Early Dry protocol — After meeting eligibility criteria, patients have a net ultrafiltration of 2mL/kg/h with systematic perfusion monitoring (lactate concentration, central venous saturation, mottling score and capillary refill time) and restrictive input.
  If the patient presents hypoperfusion (at least to sign), net ultrafiltration is stopped and haemodynamic optimized.
  If the patient presents pulmonary oedema or right ventricular failure, with venous congestion, ultrafiltration is set at 3mL/kg/h.
  Ultrafiltration is set between 0.5 and 1mL/kg/h when the following criteria are fulfilled: weight inferior to the admission weight; central venous pressure inferior to 5mmHg; absence of clinical oedema.
  The haemodynamic status is reevaluated all six hours.

SUMMARY:
Fluid overload is frequent and associated with mortality in critically ill patients, especially those with acute kidney injury. If fluid loading is a cornerstone of a resuscitation strategy, some authors promote an evacuation phase to limit the fluid overload exposure (deresuscitation strategy). In patients with continuous renal therapy, often presenting an inadequate diuresis, it includes the net ultrafiltration setting. A potential side effect of deresuscitation strategy is to induce iatrogenic hypovolemia.

We have implemented a perfusion-based protocol to induce systematic early fluid removal on patients after haemodynamic stabilization. We would like to observe the impact on the fluid balance of such a protocol and to explore the recruitment capacity of our centre and exploratory outcomes to lead a future randomized control study.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 ans
* Acute kidney injury with continuous renal replacement therapy
* Fluid overload > 5%
* Equivalent Norepinephrine dose < 0,5 µg/kg/min

Exclusion Criteria:

* - Chronic intermittent haemodialysis
* Active bleeding
* Stroke with coma
* Pregnancy
* advanced directives to withhold or withdraw life-sustaining treatment
* patient's opposition to the use of his/her personal health data."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients in intensive care unit with acute kidney injury with continuous renal replacement therapy and fluid overload, with hemodynamic instability
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Computed cumulative fluid balance (mL) at day 5 after protocol onset. | Day 5 after protocol onset.
  Cumulative between input and output, defined as follow:
  * Input = cumulative volume of:
    * Medication
    * Enteral and parenteral feeding
    * Fluid loading
    * Transfusion products
  * Output = cumulative volume of:
    * diuresis
    * surgical drainage
    * net ultrafiltration

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital cardiologique Louis Pradel - HCL, Bron, France